CLINICAL TRIAL: NCT01811004
Title: Evaluation of 1440nm Laser vs. Botulinum Toxin or miraDry® Microwave For Treatment of Axillary Hyperhidrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CYN12-GS-HH01
Record Dates: First submitted 2012-12-06; First posted 2013-03-14 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-12

CONDITIONS: Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Botox® (Experimental): Botox®
  Interventions: Device: Nd:YAG Laser; Device: Botox®
- miraDry® (Experimental): miraDry®
  Interventions: Device: miraDry; Device: Nd:YAG Laser
- Nd: YAG laser (Experimental): Nd: YAG laser 1440nm
  Interventions: Device: Nd:YAG Laser

INTERVENTIONS:
Device: miraDry — miraDry
  Arms: miraDry®
Device: Nd:YAG Laser — Nd:YAG 1440 nm Laser
Device: Botox® — Botox®
  Arms: Botox®

SUMMARY:
The Purpose of the study is to evaluate the 1440nm Laser Assisted Selective Photothermolysis vs. Botulinum Toxin or miraDry® Microwave Thermolysis For Treatment of Axillary Hyperhidrosis.

ELIGIBILITY:
Inclusion Criteria:

* A healthy non-smoking male or female between 18-70 years of age
* Understand/accept obligation not to receive any other procedures in anatomical areas exhibiting axillary hyperhidrosis through 3 months prior to treatment
* Understand and accept the obligation and is logistically able to present for all scheduled follow-up visits
* Clinically diagnosed for primary hyperhidrosis of the axilla.
* A self-assessed Hyperhidrosis Disease Severity Scale (HDSS) score of three (3) or four (4) a. Gravimetric >50mg/5min in each axilla

Exclusion Criteria:

* Clinical diagnosis of secondary hyperhidrosis
* Uncontrolled systemic disease or infection
* Concurrent use of any hyperhidrosis treatments other than over the counter antiperspirants or deodorants
* Receipt of Botox® or Dysport® within the past six months
* Patients who refuse to stop using over the counter antiperspirants 24 hours prior to the day of surgery and each of the follow-up visits at 3 months and 6 months that Minors starch iodine tests may be performed.
* Patients using or having used within 7 days of baseline visit: cholinomimetic agents, anticholinergic agents, prescription antiperspirants, any herbal medicine treatments or any other treatments for hyperhidrosis except OTC antiperspirant or planning to use such agents during the course of the study.
* Any previous liposuction/liposculpture or any type of surgery for hyperhidrosis; OR any other types of treatments for hyperhidrosis in the area to be treated in the past 6 months
* Has any other medical condition, that, in the investigator's opinion would interfere with the subject's participation in the study
* Is susceptible to light induced seizures or history of seizures
* Has a history of keloid formation
* Significant cardiovascular disease
* Bleeding disorders
* Anti-platelet and anticoagulant medication
* Sensitivity to lidocaine or epinephrine
* Pregnancy or planned pregnancy
* Existing neuromuscular disorders (myasthenia gravis, Eaton-Lambert Syndrome, amyotrophic lateral sclerosis)
* Electronic implants
* Subjects requiring supplemental oxygen
* Has therapies or medications which may interfere with the treatment (including medications causing photosensitivity
* Allergic to Keflex

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- Sasaki Advanced Aesthetic Medical Center, Pasadena, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Nd: YAG Laser and miraDry: Nd: YAG laser 1440nm and miraDry
  For each patient, one axilla was treated with the 1440 nm Diode laser and the opposite axilla was treated with miraDry. The subject is treated with miraDry at day 0, and again at day 90.
  Nd:YAG Laser: Nd:YAG 1440 nm Diode Laser with a Rep Rate of 25 Hz. Total energy around 1500 J per 5cm x 5cm sector.
- Nd: YAG Laser 1440nm and Botox: Nd: YAG laser 1440nm and Botox
  For each patient, one axilla was treated with the 1440 nm Diode laser and the opposite axilla was treated with Botox.
  Nd:YAG Laser: Nd:YAG 1440 nm Diode Laser with a Rep Rate of 25 Hz. Total energy around 1500 J per 5cm x 5cm sector.
Period: Overall Study
Arm/Group | Nd: YAG Laser and miraDry | Nd: YAG Laser 1440nm and Botox
Started | 9 | 8
Completed | 8 | 5
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Nd: YAG Laser- miraDry: Nd: YAG laser 1440nm
  miraDry: miraDry
- Nd: YAG Laser- Botox: Nd:YAG Laser: Nd:YAG 1440 nm Laser
  Botox®: Botox®
- Total: Total of all reporting groups
Arm/Group | Nd: YAG Laser- miraDry | Nd: YAG Laser- Botox | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 5 | 3 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 3 | 5 | 8
  Race/Ethnicity: Hispanic | 0 | 2 | 2
  Race/Ethnicity: Asian | 2 | 0 | 2
  Race/Ethnicity: African American | 2 | 0 | 2
  Race/Ethnicity: Puerto Rican/Caucasian | 1 | 0 | 1
  Race/Ethnicity: African American/Caucasian | 1 | 0 | 1
  Race/Ethnicity: Other (Not Specified) | 0 | 1 | 1
Fitzpatrick Skin Score [Count of Participants; unit: Participants] — The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is.
  The scale comes from this source:
  Gupta, Sharma. Skin typing: Fitzpatrick grading and others. Clinics in Dermatology. 2019;37(5):430-436. doi:10.1016/j.clindermatol.2019.07.010
  Participants
    Fitzpatrick Skin Score I | 1 | 0 | 1
    Fitzpatrick Skin Score II | 1 | 3 | 4
    Fitzpatrick Skin Score III | 1 | 3 | 4
    Fitzpatrick Skin Score IV | 4 | 2 | 6
    Fitzpatrick Skin Score V | 2 | 0 | 2
    Fitzpatrick Skin Score VI | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Sweating Assessed Using Gravimetry
Description: A gravimetry test was performed to determine the quantity of sweat produced, comparing the post-treatment to the baseline numbers. A pre-weighted filter paper was placed on the armpit, and then weighed afterwards to determine the quantity of sweat produced.
Time Frame: 1 month follow up
Population: One subject in the Botox treatment was a no-show to their scheduled follow up.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Botox® | miraDry® | Nd: YAG Laser
Number analyzed (Participants) | 7 | 9 | 16
mg | 267.91 (432.53) | 57.36 (33.55) | 155.14 (263.53)

2. Primary Outcome: Change in Sweating Assessed Using Gravimetry
Description: as for outcome 1
Time Frame: 3 month follow up
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Botox® | miraDry® | Nd: YAG Laser
Number analyzed (Participants) | 8 | 9 | 17
mg | 231.89 (407.42) | 53.59 (38.67) | 22.72 (31.34)

3. Primary Outcome: Change in Sweating Assessed Using Gravimetry
Description: as for outcome 1
Time Frame: 6 month follow up
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Botox® | miraDry® | Nd: YAG Laser
Number analyzed (Participants) | 8 | 9 | 17
mg | 223.51 (380.18) | 65.93 (46.48) | 39.07 (42.11)

4. Primary Outcome: Change in Sweating Assessed Using Gravimetry
Description: as for outcome 1
Time Frame: 9 month follow up
Population: The gravimetric test was not required for the 9 month follow up.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Botox® | miraDry® | Nd: YAG Laser
Number analyzed (Participants) | 4 | 8 | 12
mg | 99.49 (81.27) | 67.06 (44.3) | 28.36 (37.84)

ADVERSE EVENTS:
Time Frame: Adverse Events occurring were collected throughout the study, around 18 months.
Groups:
- Botox®: Botox® and Nd:YAG Laser: 1440 nm Laser
- miraDry®: miraDry® and Nd:YAG 1440 nm Laser
- Nd: YAG Laser: Nd: YAG laser: 1440nm
Arm/Group | Botox® | miraDry® | Nd: YAG Laser
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/17
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9 | 17/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botox® (N=8) | miraDry® (N=9) | Nd: YAG Laser (N=17)
Numbness (Skin and subcutaneous tissue disorders) | 7 | 9 | 16
Pain (Nervous system disorders) | 8 | 9 | 17
Redness (Skin and subcutaneous tissue disorders) | 7 | 9 | 15
Swelling (Skin and subcutaneous tissue disorders) | 8 | 9 | 15
Bruising (Skin and subcutaneous tissue disorders) | 2 | 9 | 16
Itching (Skin and subcutaneous tissue disorders) | 5 | 5 | 10
Nodule (Skin and subcutaneous tissue disorders) | 7 | 9 | 13
Hardness (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.